CLINICAL TRIAL: NCT04331899
Title: A Phase 2 Randomized, Single-Blind Study of a Single Dose of Peginterferon Lambda-1a (Lambda) Compared With Placebo in Outpatients With Mild COVID-19
Brief Title: Single-Blind Study of a Single Dose of Peginterferon Lambda-1a Compared With Placebo in Outpatients With Mild COVID-19
Acronym: COVID-Lambda
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 55619
Record Dates: First submitted 2020-03-27; First posted 2020-04-02 (Actual); Results first posted 2021-04-22 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
Keywords: Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — peginterferon lambda-1a

STUDY DESIGN:
Intervention Model Description: An open-label, single-blind randomized controlled trial. Study participants will be randomly assigned 1:1 to a single subcutaneous dose of Peginterferon Lambda-1a or placebo along with the standard of care.
Who Masked: Participant
Masking Description: Single-blind study in which only patients are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study drug Peginterferon Lambda-1a (Experimental): Study participants assigned to study drug will receive a single subcutaneous dose of Peginterferon Lambda-1a in addition to standard of care treatment.
  Interventions: Drug: Peginterferon Lambda-1a
- Placebo injection (Placebo Comparator): Study participants will receive a placebo along with the standard of care treatment.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Peginterferon Lambda-1a — Peginterferon Lambda-1a (180 ug subcutaneous injection) single dose along with Standard of Care
  Arms: Study drug Peginterferon Lambda-1a
Other: Placebo — Placebo subcutaneous injection along with Standard of Care Treatment for COVID-19 Infection
  Arms: Placebo injection

SUMMARY:
To evaluate the efficacy of a single dose of subcutaneous injections of 180 ug of Peginterferon Lambda-1a, compared with placebo in reducing the duration of viral shedding of SARS-CoV-2 virus in patients with uncomplicated COVID-19 disease.

DETAILED DESCRIPTION:
Patients will attend up to 9 study visits over a period of up to 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 75 years at the time of the assessment
2. Able and willing to understand the study, adhere to all study procedures, and provide written informed consent
3. Diagnosis of COVID-19 disease:

   1. If symptomatic, the presence of mild to moderate symptoms without signs of respiratory distress, with FDA-cleared molecular diagnostic assay positive for SARS-CoV-2 within 72 hours from swab to the time of commencing informed consent:
   2. If asymptomatic, initial diagnosis of SARS-CoV-2 infection with positive FDA-cleared molecular diagnostic assay obtained no more than 72 hours from initial swab to the time of commencing informed consent

Exclusion Criteria:

1. Patients who are hospitalized for inpatient treatment or currently being evaluated for potential hospitalization at the time of initiation of informed consent
2. Patients with a known allergy to Peginterferon Lambda-1a or any component thereof
3. Display symptoms of respiratory distress (Respiratory rate >20, room air oxygen saturation of <94%.)
4. Participation in a clinical trial with or use of any investigational agent within 30 days before screening
5. Treatment with interferons (IFN) within 12 months before screening
6. Previous use of Peginterferon Lambda-1a
7. History or evidence of any intolerance or hypersensitivity to IFNs or other substances contained in the study medication.
8. Female patients who are pregnant or breastfeeding. Male patients must confirm that their female sexual partners are not pregnant.
9. Current or previous history of decompensated liver disease (Child-Pugh Class B or C) or hepatocellular carcinoma
10. Co-infected with human immunodeficiency virus (HIV)
11. Significant abnormal laboratory test results at screening.
12. Other significant medical condition that may require intervention during the study
13. Concurrent use of any of the following medications:

    1. Therapy with an immunomodulatory agent
    2. Current use of heparin or Coumadin
    3. Received blood products within 30 days before study randomization
    4. Use of hematologic growth factors within 30 days before study randomization
    5. Systemic antibiotics, antifungals, or antivirals for treatment of active infection within 24 hours before study randomization
    6. Any prescription or herbal product that is not approved by the investigator
    7. Long-term treatment (> 2 weeks) with agents that have a high risk for nephrotoxicity or hepatotoxicity unless it is approved by the medical monitor
    8. Receipt of systemic immunosuppressive therapy within 3 months before screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-04-25 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2021-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Upinder Singh, Principal Investigator — Professor (Medicine-Infectious Diseases)
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing of generated and analyzed datasets.
Supporting Information: Study Protocol, SAP
Time Frame: The datasets generated and analyzed during the current study are permanently available in the Stanford Digital Repository
Access Criteria: Full access
URL: https://purl.stanford.edu/hc972ys6733

REFERENCES:
- [Result] Jagannathan P, Andrews JR, Bonilla H, Hedlin H, Jacobson KB, Balasubramanian V, Purington N, Kamble S, de Vries CR, Quintero O, Feng K, Ley C, Winslow D, Newberry J, Edwards K, Hislop C, Choong I, Maldonado Y, Glenn J, Bhatt A, Blish C, Wang T, Khosla C, Pinsky BA, Desai M, Parsonnet J, Singh U. Peginterferon Lambda-1a for treatment of outpatients with uncomplicated COVID-19: a randomized placebo-controlled trial. Nat Commun. 2021 Mar 30;12(1):1967. doi: 10.1038/s41467-021-22177-1. PMID 33785743
- [Derived] McCarthy MW. Interferon lambda as a potential treatment for COVID-19. Expert Opin Biol Ther. 2023 May;23(5):389-394. doi: 10.1080/14712598.2023.2211709. Epub 2023 May 8. PMID 37147857
- [Derived] van der Ploeg K, Kirosingh AS, Mori DAM, Chakraborty S, Hu Z, Sievers BL, Jacobson KB, Bonilla H, Parsonnet J, Andrews JR, Press KD, Ty MC, Ruiz-Betancourt DR, de la Parte L, Tan GS, Blish CA, Takahashi S, Rodriguez-Barraquer I, Greenhouse B, Singh U, Wang TT, Jagannathan P. TNF-alpha+ CD4+ T cells dominate the SARS-CoV-2 specific T cell response in COVID-19 outpatients and are associated with durable antibodies. Cell Rep Med. 2022 Jun 21;3(6):100640. doi: 10.1016/j.xcrm.2022.100640. Epub 2022 May 3. PMID 35588734
- [Derived] Jacobson KB, Rao M, Bonilla H, Subramanian A, Hack I, Madrigal M, Singh U, Jagannathan P, Grant P. Patients With Uncomplicated Coronavirus Disease 2019 (COVID-19) Have Long-Term Persistent Symptoms and Functional Impairment Similar to Patients with Severe COVID-19: A Cautionary Tale During a Global Pandemic. Clin Infect Dis. 2021 Aug 2;73(3):e826-e829. doi: 10.1093/cid/ciab103. PMID 33624010

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment opened on April 24, 2020. The first patient was enrolled on April 25, 2020, and the last patient was enrolled on July 17, 2020.
Groups:
- Lambda: Peginterferon Lambda-1a (Lambda) single dose administered subcutaneously in addition to standard of care treatment.
- Placebo: Placebo to match Lambda single dose administered subcutaneously in addition to standard of care treatment.
Period: Trial Period (28 Days)
Arm/Group | Lambda | Placebo
Started | 60 | 60
Completed | 58 | 58
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2
Period: Follow-up Period (10 Months)
Arm/Group | Lambda | Placebo
Started | 42 (16 participants who completed the trial period did not continue in the follow-up period.) | 43 (15 participants who completed the trial period did not continue in the follow-up period.)
Completed | 42 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lambda: Lambda single dose administered subcutaneously in addition to standard of care treatment.
- Total: Total of all reporting groups
Arm/Group | Lambda | Placebo | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Median (Full Range); unit: years] | 37 [18 to 66] | 34 [20 to 71] | 36 [18 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 50
  Male | 36 | 34 | 70
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Latinx | 34 | 41 | 75
  White | 18 | 15 | 33
  Asian | 3 | 4 | 7
  Native Hawaiian or other Pacific Islander | 2 | 0 | 2
  Unknown | 2 | 0 | 2
  More than one race | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60 | 60 | 120
Duration of symptoms prior to randomization [Median (Inter-Quartile Range); unit: days] | 4 [3 to 6] | 5 [3 to 5] | 5 [3 to 9]
Asymptomatic at baseline [Count of Participants; unit: Participants] | 6 | 2 | 8
Symptoms at baseline [Count of Participants; unit: Participants]
  Fatigue | 33 | 42 | 75
  Cough | 33 | 36 | 69
  Headache | 29 | 36 | 65
  Myalgias | 29 | 34 | 63
  Decreased taste or smell | 25 | 32 | 57
  Chills | 22 | 27 | 49
  Sore throat | 22 | 23 | 45
  Joint pain | 19 | 19 | 38
  Diarrhea | 16 | 18 | 34
  Nausea | 11 | 23 | 34
  Shortness of breath | 16 | 16 | 32
  Chest pain/pressure | 14 | 13 | 27
  Runny nose | 10 | 16 | 26
  Abdominal pain | 7 | 7 | 14
  Rash | 4 | 5 | 9
  Vomiting | 1 | 5 | 6
Body temperature ≥99.5°F [Count of Participants; unit: Participants] | 6 | 7 | 13
Oxygen saturation [Median (Inter-Quartile Range); unit: percentage of peripheral capillary O2] | 98 [97 to 100] | 99 [97 to 99.5] | 98 [97 to 100]
White blood cell count [Median (Inter-Quartile Range); unit: cells/μl] | 5.5 [4.3 to 6.8] | 5.6 [4.0 to 7.5] | 5.5 [4.1 to 7.1]
Absolute lymphocyte count [Median (Inter-Quartile Range); unit: cells/μl] | 1.5 [1.2 to 1.9] | 1.5 [1.2 to 2.3] | 1.5 [1.2 to 2.2]

OUTCOME MEASURES:

1. Primary Outcome: Duration Until Viral Shedding Cessation
Description: Time to first of two consecutive negative respiratory secretions obtained by oropharyngeal and/or anterior nare swabs for SARS-CoV-2 by qRT-PCR.
Time Frame: Assessed for up to 28 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Lambda | Placebo
Number analyzed (Participants) | 60 | 60
days | 7 [5 to 13] | 7 [5 to 10]
Statistical Analysis 1: Comparison: Lambda vs Placebo; Test type: Other; p = 0.29, Regression, Cox — Tests were conducted at the 0.05 level of significance; Cox Proportional Hazard = 0.81, 95% CI 2-sided [0.56 to 1.19] — Cox proportional hazards model covariate-adjusted for age 50+ and sex

2. Secondary Outcome: Change in Sars-CoV-2 Viral Load
Description: Log10 Oropharyngeal viral load over time, mean change at day 14 (SD). Sars-CoV-2 RNA level in oropharyngeal and/or anterior nare swabs collected daily.
Time Frame: baseline, day 14
Measure: Mean (Standard Deviation); unit: Log10 copies per mL
Arm/Group | Lambda | Placebo
Number analyzed (Participants) | 60 | 60
Log10 copies per mL | -4.3 (1.3) | -4.9 (4.7)
Statistical Analysis 1: Comparison: Lambda vs Placebo; Test type: Other; p = 0.91, Regression, Linear — Tests were conducted at the 0.05 level of significance; Cox Proportional Hazard = -0.06, 95% CI 2-sided [-1.23 to 1.11] — Log change at Day 14. Cox proportional hazards model covariate-adjusted for age 50+ and sex

3. Secondary Outcome: Area Under the Curve of SARS-COV-2 Viral Load
Description: Log10 viral load area under the curve through day 14, median (IQR). Area under the curve of SARS-CoV-2 viral load in oropharyngeal and/or anterior nare swabs collected daily.
Time Frame: baseline through day 14
Measure: Median (Inter-Quartile Range); unit: Log10 copies*days/ml
Arm/Group | Lambda | Placebo
Number analyzed (Participants) | 60 | 60
Log10 copies*days/ml | 28.5 [18.6 to 39.1] | 29.6 [19.6 to 38.7]
Statistical Analysis 1: Comparison: Lambda vs Placebo; Test type: Other; p = 0.95, Regression, Linear — Tests were conducted at the 0.05 level of significance; Cox Proportional Hazard = 1.01, 95% CI 2-sided [0.85 to 1.16] — Cox proportional hazards model covariate-adjusted for age 50+ and sex

4. Secondary Outcome: Duration Until Resolution of Symptoms
Description: Duration until resolution of symptoms in days, median (95% CI). Time to alleviation of all symptoms (fever, chills, cough, nasal congestion, muscle pains), defined as the time from initiation of treatment until all symptoms are rated as absent or mild in symptomatic patients.
Time Frame: Up to 28 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Lambda | Placebo
Number analyzed (Participants) | 60 | 60
days | 8 [6 to 11] | 9 [5 to 11]
Statistical Analysis 1: Comparison: Lambda vs Placebo; Test type: Other; p = 0.76, Regression, Cox — Tests were conducted at the 0.05 level of significance; Cox Proportional Hazard = 0.94, 95% CI 2-sided [0.60 to 1.41] — Cox proportional hazards model covariate-adjusted for age 50+ and sex

5. Secondary Outcome: Count of Participants Requiring Emergency Department Visits or Hospitalizations Within 28 Days of Initiation of Treatment
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lambda | Placebo
Number analyzed (Participants) | 60 | 60
Participants
  Hospitalizations | 2 | 2
  Emergency Department Visits | 5 | 3

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | Lambda | Placebo
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 2/60 | 2/60
Other Adverse Events (participants affected / at risk) | 15/60 | 5/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lambda (N=60) | Placebo (N=60)
Hypoxia (hospital admission) (Respiratory, thoracic and mediastinal disorders) | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lambda (N=60) | Placebo (N=60)
Elevated liver function test (Hepatobiliary disorders) | 15 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT04331899/Prot_ICF_002.pdf
  • Statistical Analysis Plan (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/99/NCT04331899/SAP_001.pdf